CLINICAL TRIAL: NCT07213466
Title: Individualized Pharmacological Approach to Obesity in Patients With Bipolar Disorder - OBOE-Mayo
Brief Title: Individualized Pharmacological Approach to Obesity in Patients With Bipolar Disorder
Acronym: OBOE-Mayo
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Mark Frye, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-005856
Record Dates: First submitted 2025-09-23; First posted 2025-10-09 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Bipolar I Disorder; Bipolar II Disorder; Schizo Affective Disorder; Obesity; Weight Loss; GLP - 1
MeSH Terms: conditions — Bipolar Disorder; Psychotic Disorders; Obesity; Weight Loss | interventions — semaglutide; Qsymia; Naltrexone-Bupropion combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Semaglutide (Wegovy) + Group Therapy Program (Experimental): By meeting the satiety/return to hunger (Hungry Gut) phenotype, participants will take Semaglutide (Wegovy) and attend a 12-week group therapy session for the 16-week clinical trial.
  Interventions: Behavioral: Group Therapy Program; Drug: semaglutide
- Naltrexone/Bupropion (Contrave) + Group Therapy Program (Experimental): By meeting the behavioral/psychological (Emotional Hunger) phenotype, participants will take Naltrexone/Bupropion (Contrave) and attend a 12-week group therapy session for the 16-week clinical trial.
  Interventions: Behavioral: Group Therapy Program; Drug: naltrexone and bupropion (combination)
- Phentermine/Topiramate (Qysmia) + Group Therapy Program (Experimental): By meeting the satiation (Hungry Brain) phenotype, participants will take Phentermine/Topiramate (Qysmia) and attend a 12-week group therapy session for the 16-week clinical trial.
  Interventions: Behavioral: Group Therapy Program; Drug: Phentermine-Topiramate
- No Study Medication + Group Therapy Program (Experimental): By meeting the slow burn phenotype, participants will attend a 12-week group therapy session for the 16-week clinical trial.
  Interventions: Behavioral: Group Therapy Program

INTERVENTIONS:
Behavioral: Group Therapy Program — a 12-week group therapy program centered around weight loss and healthy eating.
Drug: semaglutide — Brand name: Wegovy
  Arms: Semaglutide (Wegovy) + Group Therapy Program
Drug: Phentermine-Topiramate — Brand name: Qsymia
  Arms: Phentermine/Topiramate (Qysmia) + Group Therapy Program
Drug: naltrexone and bupropion (combination) — Brand name: Contrave
  Arms: Naltrexone/Bupropion (Contrave) + Group Therapy Program

SUMMARY:
The goal of this clinical trial is to identify the specific characteristics (phenotypes) that may be useful to help select the right medication for weight loss, and to study the effect of individualized guided medication in patients with bipolar disorder ages 18-65. The main questions it aims to answer are:

* Can the investigators compare the distribution of obesity characteristics (hungry brain, hungry gut, emotional hunger) between bipolar patients and non-bipolar participants (comparing from IRB #24-002375)?
* Can the investigators evaluate the feasibility of anti-obesity medication (AOM) in patients with bipolar disorder?

Participation will last for about 17-18 weeks and includes 7 in-person study visits, 4 phone call visits, and 12 virtual group therapy sessions. The first visit lasts about 2 hours and includes going over the informed consent form, a diagnostic interview to confirm diagnosis, gathering vital signs, mood questionnaires, an ECG, and urine drug and pregnancy tests (if applicable). The second visit lasts about 6-7 hours and involves multiple procedures and completing questionnaires to determine which study drug would allow participants to lose weight most effectively. At the third visit, participants will be assigned to take one of three FDA approved medications for weight loss: Semaglutide (Wegovy®), Naltrexone/Bupropion (Contrave®), or Phentermine/Topiramate (Qysmia®). It is possible that participants could be assigned to a group that receives no study medication. All participants will be enrolled in a 12-week virtual group therapy program targeted for weight loss. On this third visit the investigators will also gather vital signs, and participants will give a sample of blood. After the third visit, participants will come in for study visits every 4 weeks for 16 weeks (4 visits) to assess medication adherence, vitals, and answer questions about mood and eating (participants will also give a sample of blood at the 8-week and 16-week visits). Every two weeks in between in-person visits, the study team will call participants to assess medication adherence. Participants will be compensated for time spent in this study.

DETAILED DESCRIPTION:
This is a single-site, open-label, non-randomized interventional pilot study evaluating a phenotype-guided pharmacological approach to obesity in adults with bipolar disorder (BD). The study aims to assess the distribution of obesity phenotypes and the efficacy, safety, and tolerability of individualized anti-obesity pharmacotherapy in this population. A total of 100 participants with BD and comorbid obesity will be enrolled and stratified into one of four obesity phenotypes: Hungry Brain (abnormal satiation), Hungry Gut (abnormal postprandial satiety), Emotional Hunger (emotional eating), and Slow Burn (low resting energy expenditure).

Participants will undergo comprehensive obesity phenotyping, including indirect calorimetry, gastric emptying scintigraphy, DEXA scans, ad libitum buffet meal testing, and validated behavioral questionnaires. Based on phenotype classification, participants will receive one of the following FDA-approved anti-obesity medications (AOMs): phentermine-topiramate ER (Qsymia®), semaglutide (Wegovy®), or naltrexone-bupropion ER (Contrave®). Participants with the Slow Burn phenotype will receive behavioral and lifestyle interventions only.

All participants will engage in a 12-week virtual behavioral intervention program led by a multidisciplinary team, including a psychologist and a registered dietitian. The program includes weekly group sessions focused on nutrition, physical activity, cognitive restructuring, and relapse prevention.

A comprehensive data safety monitoring plan (DSMP) is in place, including bi-monthly reviews by a multidisciplinary team. Adverse events (AEs) and serious adverse events (SAEs) will be monitored and reported per institutional and federal guidelines. Participants will be withdrawn from the study if they experience treatment-emergent mania, severe depression, suicidality, or other safety concerns.

The statistical analysis plan includes descriptive statistics, repeated measures models, and subgroup analyses by phenotype and BD subtype. Missing data will be handled using multiple imputation or maximum likelihood methods. No formal multiplicity adjustments will be applied due to the exploratory nature of the study.

This study addresses a critical gap in obesity treatment for individuals with serious mental illness by integrating precision medicine with psychiatric care. The findings will inform future randomized controlled trials and contribute to the development of personalized obesity interventions in psychiatric populations.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between 18 to 65 years old.
* Patients with a SCID IV confirmed diagnosis of bipolar disorder (BDI or BDII) or schizoaffective bipolar type (SZA-BD).
* Women with a negative pregnancy test 48 hours before study entry (obesity phenotyping visit).
* Patients with a negative urine drug screen except for allowable drugs.
* Patients with a BMI ≥ 30 kg/m2 or a BMI ≥ 27 kg/m2 plus one medical comorbidity (e.g., type 2 diabetes, hypertension, dyslipidemia, obstructive sleep apnea)
* Patients must be undergoing mood stabilizer treatment but may also receive concurrent antidepressant or anxiolytic therapy.
* Patients must be on a stable regimen of a mood stabilizer, with no changes to the medication, for at least one month prior to study enrollment.
* Continuation of mood-stabilizing treatment is preferred but not required; the decision should be made in collaboration with the participant's primary mental health provider.

Exclusion Criteria:

* Abdominal bariatric surgery: Gastric bypass surgery (Roux-en-Y), Adjustable gastric band (Lap band), and Gastric sleeve surgery (Sleeve gastrectomy).
* Positive history of chronic gastrointestinal diseases, or systemic disease that could affect gastrointestinal motility, such as diabetic gastroparesis; or use of medications that may alter gastrointestinal motility and appetite.
* Positive history of chronic gastrointestinal diseases that could affect gastrointestinal absorption such as inflammatory bowel disease (IBD), celiac disease, small intestinal bacterial overgrowth (SIBO), etc; or use of medications that may alter gastrointestinal absorption.
* Significant untreated psychiatric dysfunction.
* Hypersensitivity to any of the study medications.
* Contraindications to the FDA-approved medications: Phentermine-Topiramate Extended Release; Oral naltrexone extended-release/bupropion extended-release (NBSR; Contrave®, Mysimba™); and Semaglutide (Weygovy™).
* Inability to provide informed consent: participants who are on involuntary commitment, conservatorship or under a legal guardian.
* Patients with active hypomania or mania (YMRS ≥ 12 points)
* Patients with active severe depression (MADRS ≥ 30 points)
* Patients with active psychosis (YMRS item 8 ≥ 6 points)
* Patients with active suicide ideation (MADRS item 10 ≥ 4 points)
* Patients with any medication changes (mood stabilizers) without advisement of study clinicians or clinical provider.
* Patients with active bulimia (purging)
* Current drug and/or alcohol use disorders (except nicotine)
* Patients with a positive toxicology screening (except cannabis)
* Positive toxicology screen for cannabis and a cannabis use disorder by CUDIT-R.
* Participants who use cannabis for recreational or medicinal purposes and fail the toxicology screen can potentially be included in the study only if they take the CUDIT-R and score a 12 or less.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Compare the distribution of obesity phenotypes (hungry brain, hungry gut, emotional hunger) between BD patients and non-BD participants (IRB #24-002375) | From enrollment through the end of the 16-week intervention.

SECONDARY OUTCOMES:
To evaluate the feasibility of anti-obesity medication (AOM) in patients with BD. | From the start of intervention (week 0) through the end of intervention (week 16).
To evaluate the tolerability of anti-obesity medication (AOM) in patients with BD. | from the start of intervention (week 0) through the end of intervention (week 16).
To evaluate changes in mitochondrial and stress-related biomarkers (e.g., MMPP metabolites and GDF15) from baseline to end point in patients with BD. | From the start of intervention (week 0) through the end of intervention (week 16).
To assess total body weight loss (in kilograms) over a 16-week period between BD patients and non-BD participants (IRB #24-002375). | From the start of intervention (week 0) through the end of intervention (week 16).
To compare the proportion of treatment responders (defined as >4% total body weight loss) over a 16-week period between BD patients and non-BD participants (IRB #24-002375). | From the start of intervention (week 0) through the end of intervention (week 16).
To evaluate changes in metabolic parameters from baseline to end point in patients with BD. | From the start of intervention (week 0) through the end of intervention (week 16).
To assess changes in eating behavior and mood symptoms from baseline to endpoint in patients with BD using validated questionnaires. | From the start of intervention (week 0) through the end of intervention (week 16).

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Frye, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No